CLINICAL TRIAL: NCT02274597
Title: Does Environmental Factors Affect Accuracy in Pre-hospital Non-invasive Temperature Measurement?
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: scs-2014
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-10

CONDITIONS: Hypothermia
Keywords: hypothermia; pre-hospital; epitympanic; temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Environmental impact on epitympanic temperature measurment: volunteers exposed to different environmental factors to simulate field settings
  Interventions: Device: metraux epitympanic thermometer

INTERVENTIONS:
Device: metraux epitympanic thermometer — accuracy of epitympanic temperature measurement in different environmental settings

SUMMARY:
The aim of this study is to assess the impact of different environmental factors on the ability for a thermistor-based epitympanic thermometer to accurately read the temperature of a normothermic individual and thereby estimate their feasibility and reliability in the austere pre-hospital setting.

DETAILED DESCRIPTION:
The aim of this study is to assess the impact of different environmental factors on the ability for a thermistor-based epitympanic thermometer to accurately read the temperature of a normothermic individual and thereby estimate their feasibility and reliability in the austere pre-hospital setting.

Healthy volunteers will be recruited. As reference value for core temperature we will use a standard rectal probe (Mon-a-Therm, General purpose Temperature Probe 12Fr/Ch, Covidien) attached to an external monitor. The study will be in a field setting in the mountains of Hemsedal, Norway.

For measuring the epitympanic temperature we will use the Metraux Thermometer (Walpoth, Galdikas et al. 1994). The Metraux Thermometer is widely used in pre-hospital care in Norway and internationally. The ear-sensor will after induction of anaesthesia be inserted according to the manufacturers specifications in the auditory canal and activated. The sensor is two tiny and soft metal wires covered in a plastic wrapping integrated in a soft rubber earplug. The depth of the measuring point is pre-set from the manufacture to be approximately 10 mm from the tympanic membrane. The display will then show the epitympanic temperature in real-time.

The volunteers will be exposed to four different scenarios. 1. Ambient air with no protection of head/measuring site. 2. Ambient air with local protection of measuring site. 3. Snow in the ear-canal before placing the thermometer (to resemble avalanche conditions). 4 Cold water in the ear canal (to resemble water immersion/submersion).

The temperature will be measured in degrees Celsius. A baseline will be established before exposing the volunteers to the different environmental factors. After exposure the temperature will be recorded every 15 seconds for a total of 10minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-60 years
* no medication
* healthy, no chronic illness
* no acute illness on study day
* No pathology in ear canal on otoscopy

Exclusion Criteria:

* Pathology in ear canal
* non-consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Temperature in degrees celsius | The patients will be followed during the induced environmental factors, an expected average of 1 hour/participant.
  The temperature will be recorded for a total of 10minutes during four different scenarios and compared to the rectal temperature

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, MD,Phd, Study Director — Division of Emergencies and Critical Care, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Skaiaa SC, Brattebo G, Assmus J, Thomassen O. The impact of environmental factors in pre-hospital thermistor-based tympanic temperature measurement: a pilot field study. Scand J Trauma Resusc Emerg Med. 2015 Sep 24;23:72. doi: 10.1186/s13049-015-0148-5. PMID 26400226